CLINICAL TRIAL: NCT06571669
Title: BOOM-IBD2 Clinical Trial to Evaluate the Effectiveness of Sacral Neuromodulation for the Treatment of IBD.
Brief Title: BOOM-IBD2 Pivotal Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boomerang Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BOOM-IBD2 (CIP-B02)
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Arm (Experimental): Patients implanted with neuromodulation
  Interventions: Device: Neuromodulation

INTERVENTIONS:
Device: Neuromodulation — Neuromodulation

SUMMARY:
The BOOM-IBD2 clinical trial is designed to evaluate the effectiveness of sacral neuromodulation for the treatment of IBD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 to 85 years of age
* Diagnosed with ulcerative colitis
* Ability and willingness to consent to participate by signing the informed consent form
* Ability to comply with the protocol and willingness to comply with all follow up requirements

Exclusion Criteria:

* Any significant medical condition that is likely to interfere with study procedures, device operation, or likely to confound the results of the study
* Any psychiatric or personality disorder at the discretion of the study investigator
* Any active bacterial infection with a risk of bacteremia or sepsis (e.g. presence of abscess)
* Active clostridium difficile infection of the colon
* Active cytomegalovirus (CMV) infection of the colon
* Evidence of colonic perforation
* Fulminant colitis requiring emergency surgery
* Microscopic, ischemic or infectious colitis
* Unresected neoplasia of the colon
* Colonic stricture unable to pass a colonoscope
* Current evidence of cancer in the gastrointestinal tract
* Current participation in another clinical trial
* Previous history of surgery for ulcerative colitis, or probably to require such intervention
* Previously implanted with a neurostimulation device or participated in a neurostimulation trial
* Inability to operate the patient programmer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Bowel Urgency | 12 weeks
  Bowel urgency at 12 weeks using the urgency numeric rating scale (URNS). The Urgency NRS is a patient-reported outcome (PRO) that quantifies the severity of bowel urgency on a scale from 0 to 10, where 0 equals no bowel urgency and 10 equals worst possible urgency.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Center for Colorectal Innovation, Los Angeles, California
  - Hoag Hospital, Newport Beach, California
  - PAMF (Palo Alto Medical Foundation), Palo Alto, California
  - Kansas Gastro, Wichita, Kansas
  - Objective Health - St. Louis, St Louis, Missouri
  - Las Vegas Medical Research LLC, DBA Vector Clinical Trials, Las Vegas, Nevada
  - Columbia University Irving Medical Center/New York Presbyterian Hospital, New York, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Objective Health - Amarillo, Amarillo, Texas
  - Objective Health - Central Texas, Waco, Texas

IPD SHARING:
Plan to Share IPD: No